CLINICAL TRIAL: NCT06079528
Title: Effect of Electromagnetic Stimulation Combined With Visceral Manipulation on Stress Urinary Incontinence In Postmenopausal Women
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Dina Mahmoud ALeshmawy Mohamed, Principal Investigator, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: DMAEMohamed
Record Dates: First submitted 2023-10-06; First posted 2023-10-12 (Actual); Last update posted 2023-10-12 (Actual); Status verified 2023-10

CONDITIONS: Stress Urinary Incontinence; Postmenopausal Disorder
MeSH Terms: conditions — Urinary Incontinence, Stress

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Electromagnetic Stimulation combined with visceral manipulation (Experimental): Consisted of 25 postmenopausal women with SUI received PEMS therapy augmented by VMT maneuvers in addition to supervised PFMT.
  Interventions: Device: Electromagnetic device; Other: visceral manipulation therapy; Other: General advice; Other: pelvic floor muscle training
- Electromagnetic Stimulation associated with general advice (Active Comparator): Control group (B) performed the same PFMT associated with general advice with no medical treatment.
  Interventions: Other: General advice; Other: pelvic floor muscle training

INTERVENTIONS:
Device: Electromagnetic device — Health wave's generator (Manufactured with Simeds S.r.l. by Machiavelli, Italy, with serial number "11492".) with two separate emission channels and asynchronous operation was employed, along with 100 saved and storable programs that could be altered by the user (intensity, frequency and phase time). The different associated applicators are recognized automatically. Magnetic field strength up to "100" Gauss and output frequency from (1 - 100) Hertz are programmable.
  Arms: Electromagnetic Stimulation combined with visceral manipulation
Other: visceral manipulation therapy — for the pelvic reproductive organs and their related structures (ligaments and fasciae) was applied one session/week for 12 weeks. Each patient was was advised to evacuate her bladder before starting the treatment session, mobility and motility testing of pelvic organs, together with the assessment of fascial tension, was then performed, with detecting restrictions, treatment was applied according to Hebgen
  Arms: Electromagnetic Stimulation combined with visceral manipulation
Other: General advice — were directed for both groups in term of the following: Perform pelvic floor exercises regularly ; avoid constipation and straining; treat the cause of any chronic cough and infection of urethra or bladder; stop smoking; maintain a healthy weight; drinking sufficient amounts of healthy fluids (water); decrease the caffeine intake; and decrease the amount of acidic and spicy foods.
Other: pelvic floor muscle training — consisted of 24 sessions of 45-60 min each, twice a week, for 12 weeks. The PFMT was divided into four phases. Proprioceptive (3 weeks): where the woman has gained adequate perception of PFM and performed fast and slow contractions; Simple (3 week): performed with the objective of promoting control of fast and slow contractions associated with small functional exercises; Elaborated (3 week): where the exercise evolved into functional exercises of greater amplitude; and Power (3 week): where the maximum voluntary contraction of the pelvic floor was promoted during efforts. In all sessions, contractions were performed for slow and fast fibers

SUMMARY:
To examine the effect of electromagnetic stimulation combined with visceral manipulation on stress urinary incontinence in postmenopausal women

DETAILED DESCRIPTION:
According to the authors' knowledge, no prior studies that included MS with a VMT maneuvers to improve the success rates of stress urinary incontinence (SUI) treatment. Consequently, the purpose of this study was to assess the effect of electromagnetic field stimulation with VMT and PFMT in treatment of postmenopausal women with SUI.

ELIGIBILITY:
Inclusion Criteria:

Fifty postmenopausal women suffering from SUI with grades mild to moderate, were referred from……..Hospital after SUI diagnosis confirmation with urodynamics. They were selected from outpatient clinic of department of physical therapy for Women's Health of the faculty of Physical Therapy, Cairo university. The inclusion criteria included sedentary and medically stable postmenopausal women, with age range of 50 to 66 years old.

Exclusion Criteria:

resence of a urinary tract infection (UTI), other types of UI, previous incontinence and pelvic floor surgeries, metallic implant, contraindications for MS, cognitive alterations, collagen or muscle-related diseases, and neurological abnormalities were exclusion criteria.

Ages: 50 Years to 66 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2022-06-01 (Actual); Primary Completion 2022-12-20 (Actual); Study Completion 2023-01-30 (Actual)

PRIMARY OUTCOMES:
Assessing the change in vaginal pressure | at baseline and after 12 weeks of intervention
  was measured by Kegel perineometer (pneumatic pelvic muscle trainer XFT-0010) designed by Shenzhen XFT Electronics co., Ltd China.

SECONDARY OUTCOMES:
Assessing the change in Urinary Incontinence symptoms | at baseline and after 12 weeks of intervention
  through the Urogenital Distress Inventory Questionnaire - Short Form (UDI-6. It is related to symptoms associated with lower urinary tract dysfunction especially SUI and it has 6 items: 1-urination frequency, 2-Leakage associated with feeling of urgency, 3-Leakage associated with activity, 4-Sneezing or Coughing little amounts of urine, 5-Emptying bladder with difficulty, and 6-Discomfort in the genital area or lower abdomen. Obtain the mean values of all the answered items then multiply by 25. Scores are turned to a possible range of 0-100. Higher scores mean more symptom distress. An "A-grade" recommendation was given to this scale by the International Consultation of Incontinence because of published data indicated that the scale is valid, reliable, and responsive to change following standard psychometric testing

CONTACTS AND LOCATIONS:
Overall Officials: Dina Mohamed, Principal Investigator — Cairo University
Locations (1):
- Outpatient clinic faculty of physical therapy cairo university, Dokki, Egypt

IPD SHARING:
Plan to Share IPD: Undecided